CLINICAL TRIAL: NCT02529787
Title: Comparative Open-label,Randomized, Fasting, Single Dose, Two-way Crossover Bioequivalence Study of Dexlansoprazole From Doxirazole 60 mg Capsules (Hikma Pharma,Egypt)and Dexilant 60 mg DR Capsules (Takeda Pharmaceuticals America Inc., USA)
Brief Title: A Bioequivalence Study of Dexlansoprazole From Doxirazole 60 mg Capsules (Hikma Pharma,Egypt)and Dexilant 60 mg Delayed Release (DR) Capsules (Takeda Pharmaceuticals America Inc., USA)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genuine Research Center, Egypt (Industry)
Collaborators: Hikma Pharma,Egypt (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: GRC/1/12/406
Record Dates: First submitted 2015-08-19; First posted 2015-08-20 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: Healthy
MeSH Terms: interventions — Dexlansoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A Test (Experimental): Test drug (Doxirazole) 1 capsule contains 60 mg of Dexlansoprazole
  Interventions: Drug: Doxirazole
- B Reference (Active Comparator): Reference drug (Dexilant) 1 capsule contains 60 mg of Dexlansoprazole
  Interventions: Drug: Dexilant

INTERVENTIONS:
Drug: Doxirazole — 1 capsule contains 60 mg Dexlansoprazole
  Other Names: Dexilant
  Arms: A Test
Drug: Dexilant — 1 capsule contains 60 mg Dexlansoprazole
  Arms: B Reference

SUMMARY:
Comparative randomized, single dose, two-way crossover open-label study to determine the bioequivalence of Dexlansoprazole from Doxirazole 60 mg Capsules (Hikma Pharma,Egypt)and Dexilant 60 mg Delayed release Capsules (Takeda Pharmaceuticals America Inc., USA)

DETAILED DESCRIPTION:
Primary Pharmacokinetic Parameters: Cmax, Area under cover (AUC0→t and AUC0→∞ ) Secondary Pharmacokinetic Parameters: Ke, tmax and t1/2e. ANOVA using 5% significance level for transformed (with the 90% confidence intervals) and untransformed data of Cmax, AUC0→t and AUC0→∞ and for untransformed data of Ke, tmax and t1/2e. The confidence intervals of logarithmically transformed Test/Reference ratios for Cmax, AUC0→t and AUC0→∞ to be within 80.00-125.00%.

A comprehensive final report will be issued upon the completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* 1. Healthy male or female, age 18 to 55 years, inclusive. 2. Body weight within 15% of normal range according to the accepted normal values for body mass index (BMI).

  3. Medical demographics without evidence of clinically significant deviation from normal medical condition.

  4. Results of clinical laboratory test are within the normal range or with a deviation that is not considered clinically significant by principal investigator.

  5. Subject does not have allergy to the drugs under investigation.

Exclusion Criteria:

* 1. Subjects with known allergy to the products tested. 2. Subjects whose values of BMI were outside the accepted normal ranges. 3. Female subjects who were pregnant, nursing or taking birth control pills. 4. Medical demographics with evidence of clinically significant deviation from normal medical condition.

  5. Results of laboratory tests which are clinically significant. 6. Acute infection within one week preceding first study drug administration. 7. History of drug or alcohol abuse. 8. Subject does not agree not to take any prescription or non-prescription drugs within two weeks before first study drug administration and until the end of the study.

  9. Subject is on a special diet (for example subject is vegetarian). 10. Subject does not agree not to consume any beverages or foods containing methyl-xanthenes e.g. caffeine (coffee, tea, cola, chocolate etc.) 48 hours prior to the study administration of either study period until donating the last sample in each respective period.

  11. Subject does not agree not to consume any beverages or foods containing grapefruit 7 days prior to first study drug administration until the end of the study.

  12. Subject has a history of severe diseases which have direct impact on the study.

  13. Participation in a bioequivalence study or in a clinical study within the last 6 weeks before first study drug administration.

  14. Subject intends to be hospitalized within 3 months after first study drug administration.

  15. Subjects who, through completion of this study, would have donated more than 500 ml of blood in 7 days, or 750 ml of blood in 30 days, 1000 ml in 90 days, 1250 ml in 120 days, 1500 ml in 180 days, 2000 ml in 270 days, 2500 ml of blood in 1 year.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-02; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | Up to 12 hours post dose in each treatment period
Area under the plasma concentration versus time curve (AUC) | Up to 12 hours post dose in each treatment period

SECONDARY OUTCOMES:
Number of subjects with adverse events (AE)s | Up to 12 hours post dose in each treatment period
  Safety and tolerability parameters will include recording of AEs
Safety assessed by vital sign measurement | Up to 12 hours post dose in each treatment period
  Vital sign measurement will include blood pressure, pulse rate, respiration rate and body temperature
Measure of clinical laboratory test values to access safety and tolerability | Up to 12 hours post dose in each treatment period
  Clinical laboratory tests will include hematology, clinical chemistry and urinalysis

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elshafeey, Ph.D. Pharma, Study Director — ahmed.elshafeey@grc-me.com
Locations (1):
- Genuine Research Center GRC, Cairo, Egypt

REFERENCES:
- [Background] Chow SC, Wang H. On sample size calculation in bioequivalence trials. J Pharmacokinet Pharmacodyn. 2001 Apr;28(2):155-69. doi: 10.1023/a:1011503032353. PMID 11381568
- [Background] Diletti E, Hauschke D, Steinijans VW. Sample size determination for bioequivalence assessment by means of confidence intervals. Int J Clin Pharmacol Ther Toxicol. 1991 Jan;29(1):1-8. PMID 2004861
- [Background] Schuirmann DJ. A comparison of the two one-sided tests procedure and the power approach for assessing the equivalence of average bioavailability. J Pharmacokinet Biopharm. 1987 Dec;15(6):657-80. doi: 10.1007/BF01068419. PMID 3450848
- See also: Description: Note for Guidance on Good Clinical Practice (CPMP/ICH/135/95) The European Agency for the Evaluation of Medicinal Products (EMEA) May 1997 — http://www.ema.europa.eu
- See also: Note for Guidance on Clinical Safety Data Management; Definitions And Standards for Expedited Reporting (CPMP/ICH/377/95) The European Agency for the Evaluation of Medicinal Products (EMEA) June 1995. — http://www.ema.europa.eu
- See also: International conference of Harmonization (ICH) of Technical Requirements for Registration of Pharmaceuticals for Human Use. ICH Harmonized Tripartite Guideline. Guidelines for Validation of Analytical Procedures: Methodology. November, 1996 — http://www.pharmaweb.net/pwmirror/pw9/ifpma/ICH1.html